CLINICAL TRIAL: NCT06695039
Title: A Phase 2, Open-label, Non-randomized, Single Center Study to Explore Diagnostic Performance of [18F]Fluoroestradiol (FES) Positron Emission Tomography/Computed Tomography for the Assessment of Axillary Lymph Node Metastasis in Estrogen-positive Breast Cancer
Brief Title: Diagnostic Performance of [18F]FES PET/CT for Axillary LN Metastasis in ER-positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sangwon Han, Clinical assistant professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FES axilla
Record Dates: First submitted 2024-09-24; First posted 2024-11-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Invasive
Keywords: breast caner; estrogen receptor; [18F]FES PET/CT; axillary lymph node

STUDY DESIGN:
Intervention Model Description: A phase 2, open-label, non-randomized, single center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]FES PET/CT (Experimental)
  Interventions: Diagnostic Test: Fluoroestradiol (18F)

INTERVENTIONS:
Diagnostic Test: Fluoroestradiol (18F) — images for 90 minutes after F-18 FES injection

SUMMARY:
This study aims to explore the diagnostic performance of [18F]FES PET/CT for the evaluation of axillary lymph node metastasis in patients with ER-positive breast cancer having clinically suspected or confirmed axillary lymph node metastasis.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among women, with around 310,000 new cases expected in the U.S. in 2024, accounting for 32% of all cancers diagnosed in women. About 75% of breast cancers express estrogen receptors (ER) at the time of diagnosis, and the axillary lymph nodes are the most common site for metastasis. Around 34% of breast cancer patients present with lymph node metastasis, with 24% classified as pN1 (1-3 lymph nodes) and 10% as pN2 or higher (4 or more lymph nodes) according to the AJCC staging system. The presence and extent of lymph node metastasis are critical in determining the stage of breast cancer, as well as predicting the likelihood of recurrence and survival after surgery. Lymph node involvement also guides decisions about the scope of surgery and systemic therapy.

To minimize complications such as lymphedema, axillary lymph node dissection (ALND) has become less invasive over time. The ACOSOG Z0011 trial demonstrated that patients with 1-2 lymph node metastases detected via sentinel node biopsy (SNB), who had no clinically evident axillary lymph node metastasis, could avoid ALND without negatively affecting their prognosis. As a result, preoperative evaluation of axillary lymph node metastasis has become increasingly important in determining the appropriate surgical approach. For systemic treatment, the NCCN guidelines recommend adjuvant chemotherapy for estrogen receptor-positive, HER2-negative breast cancer patients with pN2 or higher lymph node involvement after surgery. In cases of pN1 or pN0 (with tumors larger than 0.5 cm), the decision to administer adjuvant chemotherapy is based on the recurrence risk score from a 21-gene assay.

[18F]FES PET/CT has recently gained attention as an imaging modality for breast cancer due to its ability to evaluate ER status with high concordance to immunohistochemistry and detect metastasis. The NCCN guidelines now recommend its use in cases of recurrent or metastatic ER-positive breast cancer. In our previous research, [18F]FES PET/CT has a sensitivity of 77% and specificity of 100% for breast cancer diagnosis when compared to histopathological findings. Although its accuracy for detecting axillary lymph node metastasis specifically has not been thoroughly studied, it has shown potential in identifying difficult-to-detect axillary metastases. In one study, the use of [18F]FES PET/CT led to changes in treatment plans for about 26% of patients, particularly by identifying lymph node metastases that were missed by standard imaging techniques.

In addition to its use in recurrent or metastatic breast cancer, [18F]FES PET/CT is being investigated for its utility in evaluating axillary lymph nodes and staging early breast cancer. Preliminary studies at our hospital on invasive lobular breast cancer patients have shown that [18F]FES PET/CT has favorable diagnostic accuracy for detecting axillary lymph node metastasis. While PET resolution limits its ability to assess micrometastases, the high specificity and positive predictive value suggest that it could accurately predict the presence and burden of axillary lymph node metastasis in estrogen receptor-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 19 years or older regardless of race/ethnicity.
* Subjects with histologically confirmed moderate-to-strong estrogen receptor-positive invasive breast cancer within 90 days prior to [18F]FES PET/CT imaging
* Subjects whose primary tumor of cT1-3 according to the American Joint Committee on Cancer (AJCC) 8th tumor staging system
* Subjects with suspected or confirmed axillary lymph node metastasis clinically or in imaging test (ultrasound)
* Subjects who scheduled to undergo sentinel node biopsy or axillary lymph node dissection within 90 days of [18F]FES PET/CT imaging
* Subjects whose Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 2 points or less

Exclusion Criteria:

* Subject or the subject's legally acceptable representative does not provide written informed consent form
* Subjects with confirmed or suspected distant metastases.
* Previous history of ipsilateral axillary lymph node dissection, sentinel lymph node surgery, or lymph node dissection biopsy.
* Patients who are scheduled for or have undergone chemotherapy, radiotherapy, antihormone therapy, targeted therapy, or immunotherapy between [18F]FES PET/CT and pathological diagnosis
* Subjects who are pregnant or lactating. Exclusion of the possibility of pregnancy is made by one of the following: 1) Physiologically menopausal (menstruation has stopped for more than 2 years), 2) Surgically infertility (with a history of bilateral oophorectomy or hysterectomy), 3) In the case of subjects with a possibility of pregnancy, negative serum or urine pregnancy test before administration of [18F]FES has to be negative within 24 hours, and the subjects are instructed to use contraception during her participation in this study.
* Subject has concurrent severe and/or uncontrolled and/or unstable medical condition other than cancer (e.g., congestive heart failure, acute myocardial infarction, severe lung disease, chronic kidney disease or chronic liver disease).
* Subject is a relative or student of the investigator or otherwise in a dependent relationship
* Subject has already participated in this study
* Subject not being able to provide intact data for this study due to personal circumstances or other reasons in the judgment of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Patient based sensitivity and specificity of qualitative [18F]FES PET/CT evaluation for axillary lymph node metastasis | 80-100 minutes
  diagnostic accuracy of qualitative [18F]FES PET/CT analysis

SECONDARY OUTCOMES:
Patient based sensitivity and specificity of qualitative [18F]FES PET/CT evaluation for pN2/3 axillary lymph node metastasis | 80-100 minutes
  diagnostic accuracy of qualitative [18F]FES PET/CT analysis of pN2/3 axillary LN metastasis
Patient based sensitivity, specificity, area under ROC curve of quantitative [18F]FES PET/CT evaluation for axillary lymph node metastasis | 80-100 minutes
  diagnostic accuracy of quantitative [18F]FES PET/CT analysis
Detection rate of qualitative [18F]FES PET/CT evaluation for cN3 lymph node metastasis | 80-100 minutes
  Unexpected N3 node detection rate
Detection rate of qualitative [18F]FES PET/CT evaluation for distant metastasis | 80-100 minutes
  Unexpected M1 detection rate

CONTACTS AND LOCATIONS:
Overall Officials: Sangwon Han, Clinical assistant professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No